CLINICAL TRIAL: NCT02538120
Title: Assessment of the Neurovascular Microcirculatory Response in Diabetes Type 1
Brief Title: Assessment of the Neurovascular Microcirculatory Response in Diabetes Type 1 Patients
Acronym: NEURODIAB1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-A010008-35
Record Dates: First submitted 2015-08-14; First posted 2015-09-02 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetes type 1 patients (Active Comparator): The intervention will be : Microvascular assessment with laser speckle contrast imaging
  Interventions: Other: Microvascular assessment
- Matched control-subjects (Active Comparator): The intervention will be : Microvascular assessment with laser speckle contrast imaging
  Interventions: Other: Microvascular assessment

INTERVENTIONS:
Other: Microvascular assessment — Microvascular assessment

SUMMARY:
This study aims to see whether or not the diabetes 1 patients have a neurovascular microcirculatory dysfunction using various microvascular tests which have been previously validated.

Microvascular responses will be assessed by Laser Speckle Contrast Imaging and expressed in Laser Speckle Perfusion Units (LSPU).

DETAILED DESCRIPTION:
The investigators will compare microvascular responses between diabetes type 1 patients with matched control-subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 1 patients
* Matched control-subjects

Exclusion Criteria:

* Patients or subjects with anti-inflammatory drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Neurovascular microcirculatory response | one day
  Neurovascular response will be assessed by laser speckle contrast imaging using various microvascular tests such as deionized water iontophoresis, local heating test. Results will be explained in Laser Speckle Perfusion Units (LSPU)

CONTACTS AND LOCATIONS:
Overall Officials: Severine Dubois, MD, Principal Investigator — University Hospital
Locations (1):
- University Hospital, Angers, France

REFERENCES:
- [Derived] Marche P, Dubois S, Abraham P, Parot-Schinkel E, Gascoin L, Humeau-Heurtier A, Ducluzeau PH, Mahe G. Neurovascular microcirculatory vasodilation mediated by C-fibers and Transient receptor potential vanilloid-type-1 channels (TRPV 1) is impaired in type 1 diabetes. Sci Rep. 2017 Mar 13;7:44322. doi: 10.1038/srep44322. PMID 28287157